CLINICAL TRIAL: NCT02905851
Title: Teledermatology and Modulation of Antibiotic Dose in Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 869597
Record Dates: First submitted 2016-06-09; First posted 2016-09-19 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non Feedback (Placebo Comparator): No feedback given to this group regarding their antibiotic use Subjects take images and answer questions during the study like the feedback group, but in this group no feedback re dosing is given.
  Interventions: Other: Non Feedback group
- Feedback group (Active Comparator): Feedback given to this group regarding their antibiotic use after baseline.
  If the subject is in the feedback group, after this visit, a dermatologist will review all images and the survey results and give the patient information about whether they should:
  1. Continue current dose
  2. Reduce dose if there is at least a one point improvement in both the investigator acne global assessment AND the patient acne global assessment scores: A dose reduction will be such that the dose is halved from the previous dose. For example if the subject is on minocycline or doxycycline 100 mg twice daily, they will be reduced to minocycline or doxycycline 100 mg daily.
  3. Increase dose if had been previously reduced, dose will not be increased beyond the initial starting dose.
  Interventions: Other: Feedback group

INTERVENTIONS:
Other: Feedback group — Monitoring ability to use teledermatology to modify antibiotic burden
  Arms: Feedback group
Other: Non Feedback group — To use as control to see if antibiotic burden has been reduced in the active feedback group
  Arms: Non Feedback

SUMMARY:
To see if teledermatology can be used to reduce antibiotic burden in patients on doxycycline or minocycline for acne vulgaris

DETAILED DESCRIPTION:
The investigators are going to ascertain if antibiotic burden can be reduced with tele dermatology use.

There are two arms of the study:

1. Feedback group
2. Non feedback group

All subjects will be randomised to either group, all subjects will take photos of their face and answer questions at baseline, visit 2 (1 month), visit 3 (2 months), visit 4 (3 months).

The investigators will then use measurements of acne grading (patient grading, investigator global assessment, lesion counting, global acne grading) to reduce/taper antibiotics in the feedback group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 15 years and older
* Subjects who have been prescribed doxycycline or minocycline by their physician for acne vulgaris but have not initiated treatment yet.

Exclusion Criteria:

* Subjects who have used isotretinoin in the last 6 weeks
* Those who have used oral antibiotics within the last 4 weeks
* Those who have been initiated or changed brand of oral contraceptive pill within the last one month.
* Those subjects who cannot engage with the teledermatology platform
* Prisoners
* Adults unable to consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Reduced antibiotic use | Assessed at 4, 8, 12 weeks
  The difference in antibiotic exposure in the physician feedback group compared to those not receiving feedback

OTHER OUTCOMES:
Change in acne grading (change in patient grading) | Assessed at 4, 8, 12 weeks
  Change in Patient Grading
Change in acne grading (investigator global assessment) | Assessed at 4, 8, 12 weeks
  Change in Investigator Global Assessment
Change in acne grading (lesion counting) | Assessed at 4, 8, 12 weeks
  Change in Lesion Counting
Change in acne grading using the global acne grading | Assessed at 4, 8, 12 weeks
  Change in Global Acne Grading

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No